CLINICAL TRIAL: NCT04728659
Title: Desogestrel Versus GnRH Antagonist (Ganirelix) in IVF/ICSI Patients Undergoing Ovarian Stimulation: a Randomized Controlled Trial
Brief Title: Desogestrel Versus GnRH Antagonist in IVF/ICSI
Acronym: DEGOS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Casa di Cura Privata Villa Mafalda (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 01/2020
Record Dates: First submitted 2020-12-30; First posted 2021-01-28 (Actual); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: IVF; Infertility
Keywords: ovulation; progestin; PPOS; GnRH antagonist
MeSH Terms: conditions — Infertility | interventions — Desogestrel; ganirelix

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Desogestrel Group (Experimental): Ovulation inhibition will be performed using Desogestrel (75 mcg) starting on stimulation day 7 or when the leading follicle will reach 14 mm, whichever comes first
  Interventions: Drug: Desogestrel 0.075 MG
- GnRH antagonist (Active Comparator): Ovulation inhibition will be performed using ganirelix (Orgalutran, 0.25 mg/die) starting on stimulation day 7 or when the leading follicle will reach 14 mm, whichever comes first.
  Interventions: Drug: Orgalutran

INTERVENTIONS:
Drug: Desogestrel 0.075 MG — It will be given orally for 3 to 5 days during FSH administration for ovarian stimulation
  Arms: Desogestrel Group
Drug: Orgalutran — It will be given subcutaneously for 3 to 5 days during FSH administration for ovarian stimulation
  Arms: GnRH antagonist

SUMMARY:
Progestin primed ovarian stimulation (PPOS) has been shown to be effective in avoiding premature spontaneous ovulation, without affecting the number of retrieved oocytes or the quality of the embryos obtained. The utilization of progestins permits lower costs, an easier administration (oral assumption instead of injections) and a tight control over LH levels. Hence the PPOS may be a valid alternative to the standard ovarian stimulation protocols.

Additionally, it may be anticipated some degree of superiority of PPOS in particular categories of patients: donors, women at risk of OHSS, women who preserve their as well as poor responder or suboptimal responders for whom oocytes/embryo accumulation or double ovarian stimulation protocols are proposed The aim of this trial will be to investigate the use of Desogestrel in controlling the LH surge during ovarian stimulation in IVF/ICSI cycles. This study is a noninferiority trial in which the the primary efficacy endpoint will be the number of oocytes retrieved per patient.

Sample size calculation was performed with the assumptions that the non-inferiority margin is corresponding to three or less oocytes . With the objective to demonstrate that the difference in average number of oocytes retrieved between the Desogestrel and the ganirelix groups would not exceed three, the power for a comparison between the two groups would be equal to 87% for 75 evaluable patients in each treatment groups (for an allocation of 1:1 and a total sample size of 150). To allocate at least 150 patients, an additional 10% to cover possible dropping out were planned to allocate. A total of 165 patients will be included in this study Patients will be assigned to either the study or the control group. The study group will be administered follitropin alfa (Bemfola 150-225 IU/die) and Desogestrel (Cerazette 75 mcg daily ) will be started on stimulation day 7 or when the leading follicle will reach 14 mm, whichever comes first. An antagonist protocol will be used for the control group. Patients will be administered follitropin alfa (Bemfola 150 - 225 IU/die) and Ganirelix (Orgalutran 0.25 mg/die) will be started on stimulation day 7 or when the leading follicle will reach 14 mm, whichever comes first. When a diameter of 18 mm is reached, the final stage of oocyte maturation will be triggered with triptorelin 0.2 mg + hCG 1000 U s.c. Fertilization of the aspirated oocytes will be carried out in vitro, by either conventional insemination or ICSI, depending on semen parameters. Viable embryos will be then frozen by means of vitrificaton on the day in which they will reach the blastocyst developmental stage.

DETAILED DESCRIPTION:
Study design A prospective controlled randomized clinical trial (RCT) will be conducted to assess the non inferiority of Desogestrel (75 mcg) versus a flexible GnRH antagonist protocol with ganirelix (0.25 mg/day) in ovarian stimulation cycles.All partecipants will provide informed consent after counselling for infertility treatments and routine IVF procedures.

This will be a prospective non-inferiority trial. Given the possibility of dropouts, the study will be designed to include a total of 165 patients Patients will be recruited consecutively and allocated to one of the two groups in alternating manner.

Sample size The number of oocytes retrieved will be the primary efficacy endpoint of the study. Sample size calculation was performed with the assumptions that the non-inferiority margin is corresponding to three or less oocytes . With the objective to demonstrate that the difference in average number of oocytes retrieved between the Desogestrel and the ganirelix groups would not exceed three, the power for a comparison between the two groups would be equal to 87% for 75 evaluable patients in each treatment groups (for an allocation of 1:1 and a total sample size of 150). To allocate at least 150 patients, an additional 10% to cover possible dropping out were planned to allocate.

Ovarian stimulation Patients will be screened using transvaginal ultrasound on menstrual cycle day 2 to 3 . Patients will be then assigned to either the study or the control group. The study group will be administered follitropin alfa ( Bemfola 150 - 225 UI/die) from day 2-3 onward. The initiating dose of follitropin alfa will be decided upon the antral follicle count (AFC). After 4-5 days, ultrasound examination will be performed and the dose of FSH will be adjusted according to follicle development. Ovulation inhibition will be performed using Desogestrel (Cerazette, 75 mcg) starting on stimulation day 7 or when the leading follicle will reach 14 mm, whichever comes first. When the dominant follicles will reach 18 mm in diameter, the final stage of oocyte maturation will be triggered with triptorelin (Decapetyl) 0.2 mg s.c and serum FSH, LH, E2 and P concentrations will be measured using patients' blood tests on the same day of oocyte maturation. Transvaginal ultrasound-guided oocyte retrieval will be conducted 34 - 36 hours after trigger. All follicles with diameter of more than 10 mm will be retrieved.

An antagonist protocol will be used for the control group. Patients will be administered follitropin alfa (Bemfola 150 - 225 IU/die) from day 2-3 onward, with the dose of FSH administration based on the same criteria as for the study group. After 4-5 days, ultrasound examination will be performed and the dose of FSH will be adjusted according to follicle development. Ovulation inhibition will be performed using ganirelix (Orgalutran, 0.25 mg/die) starting on stimulation day 7 or when the leading follicle will reach 14 mm, whichever comes first. When dominant follicles reach 14 mm in diameter. When a diameter of 18 mm is reached, the final stage of oocyte maturation will be triggered with triptorelin (Decapeptyl) 0.2 mg s.c and serum FSH, LH, E2 and P concentrations will be measured using patients' blood tests on the same day of oocyte maturation.

Fertilization of the aspirated oocytes will be carried out in vitro, by either conventional insemination or ICSI, depending on semen parameters. According to the number and regularity of the blastomers and the degree of embryonic fragmentation, good-quality embryos will be frozen by means of vitrificaton on the third day after oocyte retrieval, and non-top quality embryos will placed in extended culture, out of which good morphological grade blastocysts were frozen on day 5.

ELIGIBILITY:
Inclusion Criteria:

* regular menstrual cycles over the previous 3-month period (25 - 35 days in duration)
* basal serum FSH concentration of no more than 10 IU/L

Exclusion Criteria:

* documented ovarian failure, including basal FSH above 10 IU/L or no antral follicles by ultrasound examination
* diagnosis of polycystic ovarian syndrome
* any controindication to ovarian stimulation treatment.

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 165 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-01-30 (Estimated); Study Completion 2022-02-28 (Estimated)

PRIMARY OUTCOMES:
Number of retrieved oocyte | 14 days after ovarian stimulation
  The number of retrieved oocytes after ovarian stimulation

SECONDARY OUTCOMES:
Number of patients with LH surge | During the 14 days of ovarian stimulation
  Spontaneous LH surge
cycle cancellation rate | 14 days after ovarian stimulation
  number of cancelled cycles
number of embryos | 7 days after oocyte reatrieval
  number of embryos available per couple
number of mature oocytes | 14 days after ovarian stimulation
  number of mature oocytes
serum levels of progesterone | 14 days after ovarian stimulation
  serum progesterone levels on the day of hCG

CONTACTS AND LOCATIONS:
Locations (1):
- Villa Mafalda, Roma, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] La Marca A, Capuzzo M, Sacchi S, Imbrogno MG, Spinella F, Varricchio MT, Minasi MG, Greco P, Fiorentino F, Greco E. Comparison of euploidy rates of blastocysts in women treated with progestins or GnRH antagonist to prevent the luteinizing hormone surge during ovarian stimulation. Hum Reprod. 2020 Jun 1;35(6):1325-1331. doi: 10.1093/humrep/deaa068. PMID 32395749
- [Background] Ata B, Capuzzo M, Turkgeldi E, Yildiz S, La Marca A. Progestins for pituitary suppression during ovarian stimulation for ART: a comprehensive and systematic review including meta-analyses. Hum Reprod Update. 2021 Jan 4;27(1):48-66. doi: 10.1093/humupd/dmaa040. PMID 33016316
- [Background] La Marca A, Capuzzo M. Use of progestins to inhibit spontaneous ovulation during ovarian stimulation: the beginning of a new era? Reprod Biomed Online. 2019 Aug;39(2):321-331. doi: 10.1016/j.rbmo.2019.03.212. Epub 2019 Mar 29. PMID 31138494